CLINICAL TRIAL: NCT04842617
Title: A Multicenter, Randomized, Double-blind Phase III Study：SHR6390/Placebo Combined With Endocrine Therapy for the Adjuvant Treatment of Hormone Receptor Positive,Human Epidermal Receptor 2 Negative, Node-positive, High Risk, Early Stage，Female Breast Cancer
Brief Title: Phase III Study ：SHR6390/Placebo Combined With Endocrine Therapy for the Adjuvant Treatment of Hormone Receptor Positive,Human Epidermal Receptor 2 Negative
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR6390-III-303
Record Dates: First submitted 2021-03-30; First posted 2021-04-13 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Hormone Receptor Positive,Human Epidermal Receptor 2 Negative, Node-positive, High Risk, Early Stage，Female Breast Cancer

STUDY DESIGN:
Intervention Model Description: SHR6390 Tablets compared with placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental)
  Interventions: Drug: SHR6390
- Treatment group B (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: SHR6390 — SHR6390 combined with endocrine therapy
  Arms: Treatment group A
Drug: placebo — placebo combined with endocrine therapy
  Arms: Treatment group B

SUMMARY:
The study is to evaluate the efficacy and safety of SHR6390 combined with endocrine therapy for the adjuvant treatment of hormone receptor positive,Human Epidermal Receptor 2 negative.

To observe the PK characteristics of SHR6390 combined with endocrine therapy for the adjuvant treatment of hormone receptor positive,Human Epidermal Receptor 2 negative.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal or premenopausal/perimenopausal female patients aged ≥18 years and ≤75 years old.
2. Pathological examination diagnosed as invasive breast cancer with HR+ and HER2-.
3. Underwent radical resection of breast cancer.
4. The score of ECOG was 0 - 1.
5. Fertile women must have a negative serum pregnancy test within 7 days before randomization, and be willing to use acceptable non hormonal contraceptive measures.
6. With my consent and informed consent, I am willing and able to comply with the planned visit, study treatment plan, laboratory examination and other test procedures.

Exclusion Criteria:

1. This Pathological examination diagnosed as HER2-positive breast cancer.
2. The history of any malignant tumor other than breast cancer within 5 years before randomization.
3. At the same time participate in other anti-tumor therapy clinical trials (including endocrine therapy or immunotherapy, etc.).
4. In the 6 months before randomization, the following conditions occurred: myocardial infarction, severe/unstable angina pectoris, , etc
5. Inability to swallow, intestinal obstruction, or other factors that affect the administration and absorption of the drug.
6. There are other serious physical or mental illnesses or laboratory abnormalities that may increase the risk of participating in the study, or interfere with the results of the study, as well as patients who the investigator believes are not suitable for participating in this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5274 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2031-10-31 (Estimated)

PRIMARY OUTCOMES:
IDFS（Invasive Disease-Free Survival） | at least 5 years from the date of randomization .

SECONDARY OUTCOMES:
DFS(Disease-Free Survival) | The observation time is at least 5 years from the date of randomization . Evaluations were conducted every 26 weeks for the first 2 years and every 52 weeks thereafter, with a follow-up of at least 5 years.
OS(Overall Survival) | up to approximately 5 years.
DDFS(Distant Disease-Free Survival) | from randomization to distant recurrence or death from any cause, whichever occurs first. Evaluations were conducted every 26 weeks for the first 2 years and every 52 weeks thereafter, with a follow-up of at least 5 years.
Number of Participants With adverse events (AEs) and serious adverse events (SAEs) Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v5.0. | up to approximately 5 years
  To evaluate the safety and tolerability of SHR6390 combined with endocrine therapy for the adjuvant treatment of hormone receptor positive,Human Epidermal Receptor 2 negative female breast cancer.
Plasma concentration of SHR6390 will be analyzed for PK samples | collected on day 1 of the 5th, 9th, 13th and 17th weeks, respectively.
  To explore the PK characteristics of SHR6390 combined with endocrine therapy for the adjuvant treatment of hormone receptor positive,Human Epidermal Receptor 2 negative female breast cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China